CLINICAL TRIAL: NCT00810095
Title: A Feasibility Trial to Evaluate the MindFrame System in the Recanalization of Occluded Vessels in Patients Experiencing an Ischemic Stroke
Brief Title: Percutaneous Recanalization in Ischemic Stroke Management (PRIISM): A Feasibility Clinical Study
Acronym: PRIISM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MindFrame, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-PRIISM-01
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Ischemic Stroke
Keywords: Cerebral Infarction; Stroke; Vascular Diseases; Central Nervous System Diseases; Penumbra; Functional Outcome; Aphasia; Hemiplegia; Left sided weakness; Right Sided weakness
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Stroke; Vascular Diseases; Central Nervous System Diseases; Aphasia; Hemiplegia | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: MindFrame System

INTERVENTIONS:
Device: MindFrame System — Thrombectomy Catheter designed to rapidly restore blood flow in patients experiencing an ischemic stroke
  Other Names: IRIIS System; Clot; Thrombus; Mechanical Thrombectomy; Ischemic Stroke; Intervention; Neurovascular

SUMMARY:
The primary study objective is to assess the feasibility of using the MindFrame System to safely and effectively restore blood flow in a thrombotic neurovascular occlusion in patients experiencing an ischemic stroke.

DETAILED DESCRIPTION:
The objective of PRIISM is to assess the feasibility of using the MindFrame System to safely and effectively restore blood flow in a thrombotic neurovascular occlusion in patients with acute ischemic stroke. Safety will be assessed by the device-related serious event rate as it compares to other similar therapies. The events include but are not limited to symptomatic hemorrhage, vessel dissection, embolization and overall morbidity and mortality. Target vessels include the basilar, internal carotid and middle cerebral (M1 and M2 segments) arteries.

ELIGIBILITY:
Inclusion Criteria:

1. NIHSS 6 to 30 within 6 hours of symptom onset
2. Pre-stroke Modified Rankin Score ≤ 2
3. Large Vessel Occlusion
4. Patient/patient guardian is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluation.
5. Patients must meet at least one of the following criteria:

   * Eligible for Intravenous rt-PA
   * Eligible for Intra-arterial rt-PA - IA rt-PA initiated within 6 hours of symptom onset
   * Patient presents within 6 hours of symptom onset

Exclusion Criteria:

1. Pregnancy
2. Glucose <50mg/dL
3. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR>3.0
4. Patient received heparin within 48 hours with a PTT greater than 2 times the lab normal.
5. Patient has baseline platelets < 30,000
6. Evidence of rapidly improving neurological signs of stroke at time of enrollment
7. Coma
8. Pre-existing neurological or psychiatric disease that could confound the study results
9. Known severe allergy to contrast media or nitinol
10. Patient has severe sustained hypertension
11. CT/MRI scan reveals significant mass effect with midline shift
12. Patient's angiogram shows an arterial stenosis >50% proximal to the embolus.
13. Patient's anticipated life expectancy is less than 3 months
14. Participation in another clinical investigation that could confound the evaluation of the study device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bendszus, MD, PhD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- MindFrame System Treatment Group: All participants with acute ischemic stroke who were treated with the 1st generation MindFrame System of neurothrombotic stent retrievers. The first generation MindFrame System was a self-expanding nitinol stent retriever mounted on a hypotube delivery wire and delivered to the occlusion site via a 0.027 inch microcatheter. Eligible patients were aged 18-80 years, had a baseline NIHSS score of 6-30, had a thrombotic occlusion of the ICA, MCA (M1 or M2) or basilar arteries, and could be treated within 6 hours of stroke onset.
Period: Overall Study
Arm/Group | MindFrame System Treatment Group
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: All participants treated with the Test System
Arm/Group | Treatment Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Region of Enrollment [Number; unit: participants]
  Sweden | 23
  Germany | 14
  Poland | 3
Mean Baseline National Institutes of Health Stroke Scale (NIHSS) score [Mean (Standard Deviation); unit: NIHSS units] — The NIH stroke scale (abbreviated NIHSS)is a scale developed by National Institutes of Health that communicates several different neurological deficits upon a single axis, represented by a score from 0 to 42 with "0" being no deficits and "42" being death.
  NIHSS units | 16.5 (4.7)
Median Baseline NIHSS score [Median (Full Range); unit: NIHSS units] — The NIH stroke scale (abbreviated NIHSS)is a scale developed by National Institutes of Health that communicates several different neurological deficits upon a single axis, represented by a score from 0 to 42 with "0" being no deficits and "42" being death.
  NIHSS units | 16 [8 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Technical Device Success by as Assessed by the Percentage of Participants Which Established at Least TIMI 2 Flow Upon Deployment of the System Across the Occlusion and Within 30 Minutes of Placing the Guide Catheter.
Description: TIMI Flow is a perfusion scoring system from 0-3 referring to levels of blood flow assessed during reperfusion procedures:
  TIMI 0 flow (no perfusion) TIMI 1 flow (penetration without perfusion) TIMI 2 flow (partial reperfusion) TIMI 3 flow (complete perfusion) is normal flow
Time Frame: Immediately postprocedure
Population: All participants treated with the Test System
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 40
percentage of participants | 75

2. Primary Outcome: Procedural Success as Determined by the Overal Percentage of Patients Who Achieve TIMI Grade 2/3 Flow, With or Without the Use of Adjuvant Therapy, in All Treatable Vessels as Confirmed by the Final Post Treatment Angiogram.
Description: TIMI Flow is a scoring system from 0-3 referring to levels of blood flow assessed during percutaneous coronary angioplasty:
  TIMI 0 flow (no perfusion) TIMI 1 flow (penetration without perfusion) TIMI 2 flow (partial reperfusion) TIMI 3 flow (complete perfusion) is normal flow
Time Frame: Immediately postprocedure
Population: Percentage of participants who achieved (TIMI/TICI grade 2/3 flow), with or without the use of adjuvant therapy, in all treatable vessels as confirmed by the final post treatment angiogram.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 40
percentage of participants | 82.5

3. Primary Outcome: Clinical Success
Description: Clinical Success as determined by achievment of a Modified Rankin Scale score of 0-2 at 90 days postprocedure. The modified Rankin Scale is a measure of a patient's level of functional independence with 0=normal and 6-death. Patients with a score of 0-2 are considered functionally independent.
Time Frame: 90 days postprocedure
Population: Percentage of participants achieving a Modified Rankin Scale score of 0-2 at 90 days postprocedure.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 40
percentage of participants | 47.5

4. Secondary Outcome: Number of Device-related Serious Adverse Events
Description: Evaluation of the safety of using the MindFrame System based on device-related serious adverse event(s). Device-related serious adverse events are defined as vessel perforation, intramural arterial dissection, device-related symptomatic intracranial hemorrhage, and significant embolization in a previously uninvolved arterial territory.
Time Frame: Treatment to 90 days postprocedure
Population: Per protocol analysis of all participants treated with the 1st generation MindFrame System of neurothrombotic stent retrievers.
Measure: Number; unit: events
Arm/Group | Treatment Group
Number analyzed (Participants) | 40
events | 2

ADVERSE EVENTS:
Time Frame: All adverse events up to and including the 90-day follow-up
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 12/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=40)
Intracranial hemorrhage (Nervous system disorders) | 6 (6)
Death (General disorders) | 8 (8)
Disorientation (Nervous system disorders) | 1 (2)
Malignant infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=40)
Epistaxis (Vascular disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No